CLINICAL TRIAL: NCT03424577
Title: A Randomized Phase 1 Food-Effect Study of H3B-6527 in Healthy Subjects
Brief Title: A Study to Evaluate the Food-Effect of H3B-6527
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: H3 Biomedicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H3B-6527-A001-001
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Healthy Participants
Keywords: H3B-6527; Healthy Participants; Pharmacokinetics
MeSH Terms: interventions — H3B-6527

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- H3B-6527 (Experimental): Healthy male participants will be randomly assigned to 1 of 2 possible treatment sequences: either H3B-6527 capsule with food on Day 1 and H3B-6527 capsule without food on Day 5 (treatment sequence fed/fasted), or H3B-6527 capsule without food on Day 1 and H3B-6527 capsule with food on Day 5 (treatment sequence fasted/fed).
  Interventions: Drug: H3B-6527

INTERVENTIONS:
Drug: H3B-6527 — Oral capsule

SUMMARY:
This study will be conducted to determine the effect of food on the relative bioavailability of H3B-6527 following administration of a H3B-6527 capsule with and without a meal.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy male between the ages of 18 and 55 years old
* Body mass index (BMI) >18 and ≤ 29 kilograms per meters squared (kg/m^2)
* Participants who have not had a successful vasectomy and are partners of women of childbearing potential must use a medically effective method of contraception with their partner during the study period through 30 days after the last dose of study drug. No sperm donation is allowed during the study period or for 30 days after study drug discontinuation

Exclusion Criteria:

* Participants with clinically significant heart, liver, gastrointestinal, kidney, lung, hormonal, blood, nerve or psychiatric disease or history of gastrointestinal surgery or gall bladder removal that could effect the uptake, distribution or elimination of H3B-6527
* Participants with a history of drug or alcohol misuse within 6 months prior to screening or a positive urine drug test
* Participants diagnosed with acquired immune deficiency syndrome (AIDS), or who test positive for human immunodeficiency virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV)
* Participated in another clinical trial less than 4 weeks prior to dosing or is currently enrolled in another clinical trial
* Received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within 1 week prior to the first dose
* Participants used any prescription or over-the-counter drugs within 2 weeks prior to the first dose

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Mean area under the plasma-concentration time curve from time 0 through the last measurable concentration (AUC0-t) of H3B-6527 | Days 1 and 5: Pre-dose, and 1, 2, 3, 4, 8, 12, and 16 hours postdose. Days 2 and 6: 24 and 36 hours postdose
Mean area under the plasma concentration-time of maximum observed last measurable concentration (tmax) of H3B-6527 | Days 1 and 5: Pre-dose, and 1, 2, 3, 4, 8, 12, and 16 hours postdose. Days 2 and 6: 24 and 36 hours postdose
Mean maximum observed plasma concentration (Cmax) of H3B-6527 | Days 1 and 5: Pre-dose, and 1, 2, 3, 4, 8, 12, and 16 hours postdose. Days 2 and 6: 24 and 36 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

REFERENCES:
- [Derived] Rioux N, Kim A, Nix D, Bowser T, Warmuth M, Smith PG, Schindler J. Effect of a high-fat meal on the relative bioavailability of H3B-6527, a novel FGFR4 inhibitor, in healthy volunteers. Cancer Chemother Pharmacol. 2019 Jan;83(1):91-96. doi: 10.1007/s00280-018-3708-3. Epub 2018 Oct 27. PMID 30368584